CLINICAL TRIAL: NCT00358293
Title: A Double-Blind, Randomized, Crossover Study to Evaluate the Clinical Efficacy and Safety of Oral Tizanidine HCl (12 mg) Versus Novel Sublingual Tizanidine HCl (12 mg) for the Treatment of Spasticity in MS Patients
Brief Title: Study of Nighttime Dosing of Sublingual Tizanidine (12 mg) in Multiple Sclerosis (MS) Patients With Significant Spasticity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teva GTC (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol C2/5/TZ-MS-05
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-04

CONDITIONS: Muscle Spasticity
Keywords: Multiple Sclerosis; Spasticity; Sublingual Tizanidine; Ashworth Scores; Spasticity in Multiple Sclerosis Patients
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis | interventions — tizanidine; Administration, Sublingual

INTERVENTIONS:
Drug: Tizanidine (sublingual or oral)

SUMMARY:
Nightly administration of 8 mg of a unique sublingual (under the tongue) formulation of tizanidine, a known anti-spasticity medication, has been shown in a previous study to improve next-day spasticity, about 12 hours following dosing in 20 multiple sclerosis (MS) patients. This improvement was statistically significant when compared to oral tizanidine dosing. The current study is being undertaken to see if increasing the dose to 12 mg once nightly will result in an even greater improvement, with a longer effect, i.e., next day improvement in spasticity both in the morning as well as in the late afternoon.

DETAILED DESCRIPTION:
Sublingual tizanidine, a novel test formulation of the known effective antispasticity agent, has been shown to have a unique pharmacokinetic profile [(i.e., nearly twice the bioavailability/AUC), but with little or no increase in peak plasma levels (Cmax) as compared to oral tizanidine (Zanaflex)]. When administered nightly to 20 MS patients, at a dose of 8 mg, it was shown to improve next-day spasticity (statistically significant improvement in Ashworth scores) about 12 hours post-dosing), improvement in nighttime (first quartile) sleep efficiency (as demonstrated by actigraphic measurement), and no increase in daytime somnolence.

Current study is being undertaken to evaluate if increased dosing (12 mg once nightly) of sublingual tizanidine (vs. oral) will show a concomitant increase in clinical effect, i.e., longer improvement, with next-day spasticity score improvement both in AM (as previously) as well as at PM (late afternoon) evaluation, with no increase in daytime somnolence.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 20-65
* Definitive diagnosis of MS, with Expanded Disability Status Scale (EDSS) less than 6.5 at screening
* Has significant spasticity (total Ashworth => 6) at screening
* Can maintain sleep regimens of at least 5 hours nightly for study duration
* May be allowed to take other anti-spasticity medication during study (including oral baclofen) as per individual dosing regimen, with the following qualifications:

  * No dose after 6pm on any study day
  * No dose at all on a clinic evaluation day (Visits 3, 4, 5)
* Females must agree to use a medically accepted form of birth control, be surgically sterile, or be two years post-menopausal. Oral contraception is contraindicated with tizanidine use.

Exclusion Criteria:

* Acute MS exacerbation requiring treatment with steroids within 30 days of screening
* Initiation of discontinuation of interferon beta within 30 days of screening
* Use of baclofen pump
* Use of CYP1A2 inhibitors during study
* Taking medications that would potentially interfere with the actions of the study medication or outcome variables, including: sedatives, stimulants, anti-hypertensives, tricyclic antidepressants, etc.
* Previous diagnosis of a sleep disorder, distinct from MS, such as obstructive sleep apnea or narcolepsy
* Score >18 on Beck Depression Inventory at screening
* Changes in chronic oral medications within 2 weeks of baseline and during study
* Significant abnormalities in screening lab parameters (ex: ALT, AST, bilirubin > 2 x upper limit of normal [ULN]; creatinine > 2 mg/dl; white blood cell [WBC] < 2,300; platelets < 80,000).
* Previous history of dementia, unstable psychiatric disease, or current signs and symptoms of significant medical disorders such as severe, progressive, or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, neurological, or cerebral disease
* History of allergy to tizanidine or any inactive component (including lactose intolerance) of test or reference formulation
* History of substance abuse within the past 12 months
* Within 30 days of baseline, worked a rotating or nighttime shift
* Participation in another clinical trial within 30 days of baseline
* Patients who are uncooperative or unwilling to sign consent form

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-12; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy - improvement in next-day spasticity (Ashworth scores)
Safety - no increase in next-day somnolence (measured objectively using PVT psychomotor vigilance task monitoring) and subjectively, using Epworth Sleepiness Scale (ESS) and Fatigue Severity Scale (FSS) questionnaires

SECONDARY OUTCOMES:
Secondary clinical efficacy - objective measure of sleep (actigraphy measures)

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Karni, MD, Principal Investigator — Department of Neurology, Tel Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center- Neurology Department, Tel Aviv, Israel